CLINICAL TRIAL: NCT03036852
Title: A Phase 2, Multicenter, Open-Label Study to Evaluate the Efficacy and Safety of Sofosbuvir/Velpatasvir for 12 Weeks in Subjects With Chronic HCV Infection Who Are on Dialysis for End Stage Renal Disease
Brief Title: Sofosbuvir/Velpatasvir in Adults With Chronic Hepatitis C Virus Infection Who Are on Dialysis for End Stage Renal Disease
Acronym: SOF/VEL ESRD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-342-4062; 2016-003625-42 (EudraCT Number)
Record Dates: First submitted 2017-01-27; First posted 2017-01-30 (Estimated); Results first posted 2019-11-12 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2019-11

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- SOF/VEL (Experimental): SOF/VEL for 12 weeks
  Interventions: Drug: SOF/VEL

INTERVENTIONS:
Drug: SOF/VEL — 400/100 mg fixed-dose combination (FDC) tablet(s) administered orally once daily
  Other Names: GS-7977/GS-5816; Epclusa®

SUMMARY:
The primary objectives of this study are to evaluate safety, efficacy, and tolerability of treatment with sofosbuvir/velpatasvir (SOF/VEL) for 12 weeks in adults on dialysis for end stage renal disease (ESRD) with chronic hepatitis C virus (HCV) infection of any genotype.

ELIGIBILITY:
Key Inclusion Criteria:

* Chronic HCV infected, male and non-pregnant/non-lactating females aged 18 years or older who are on dialysis for ESRD, including adults with HIV co-infection if they are suppressed on a stable, protocol-approved antiretroviral (ARV) regimen for ≥8 weeks prior to screening.

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2018-08-13 (Actual); Study Completion 2018-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (22):
- Royal Adelaide Hospital, Adelaide, South Australia, Australia
- Canada (6):
  - Kaye Edmonton Clinic, Edmonton, Alberta
  - Gordon and Leslie Diamond Health Care Center, Vancouver General Hospital, UBC Division of Gastroenterology, Vancouver, British Columbia
  - William Osler Health System- Brampton Civic Hospital, Brampton, Ontario
  - Hamilton Health Sciences - McMaster University Medical Centre Site, Hamilton, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Centre de Recherche du Centre Hospitalier de l'Universite de Montreal (CRCHUM), Montreal, Quebec
- Israel (3):
  - Shaare Zedek Medical Center, Jerusalem
  - The Chaim Sheba Medical Centre, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Auckland City Hospital, Grafton, Auckland, New Zealand
- Spain (4):
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda
  - Hospital Universitario Virgen del Rocío, Seville
- United Kingdom (7):
  - Gartnavel General Hospital, Glasgow
  - Barts Health NHS Trust, London
  - King's College Hospital, London
  - Chelsea and Westminster Hospital, London
  - Imperial College Healthcare NHS Trust, London
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

REFERENCES:
- [Result] Borgia SM, Dearden J, Lurie Y, Shafran SD, Brown A, Hyland RH, et al. Sofosbuvir/Velpatasvir for 12 Weeks Is Safe and Effective in Patients Undergoing Dialysis. American Association for the Study of Liver Diseases (AASLD); 2018 09-13 November; San Francisco, CA.
- [Derived] Borgia SM, Dearden J, Yoshida EM, Shafran SD, Brown A, Ben-Ari Z, Cramp ME, Cooper C, Foxton M, Rodriguez CF, Esteban R, Hyland R, Lu S, Kirby BJ, Meng A, Markova S, Dvory-Sobol H, Osinusi AO, Bruck R, Ampuero J, Ryder SD, Agarwal K, Fox R, Shaw D, Haider S, Willems B, Lurie Y, Calleja JL, Gane EJ. Sofosbuvir/velpatasvir for 12 weeks in hepatitis C virus-infected patients with end-stage renal disease undergoing dialysis. J Hepatol. 2019 Oct;71(4):660-665. doi: 10.1016/j.jhep.2019.05.028. Epub 2019 Jun 11. PMID 31195062

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Canada, the United Kingdom, Spain, Israel, New Zealand, and Australia. The first participant was screened on 22 March 2017. The last study visit occurred on 07 November 2018.
Pre-assignment Details: 78 participants were screened.
Groups:
- SOF/VEL: Sofosbuvir/velpatasvir (SOF/VEL) (400/100 mg) fixed-dose combination (FDC) tablet orally once daily for 12 weeks
Period: Overall Study
Arm/Group | SOF/VEL
Started | 59
Completed | 53
Not Completed | 6
Not completed — Death | 2
Not completed — Lack of Efficacy | 2
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- SOF/VEL (GT-1): SOF/VEL (400/100 mg) FDC tablet orally once daily for 12 weeks in participants with genotype 1 (GT-1) HCV infection
- SOF/VEL (GT-2): SOF/VEL (400/100 mg) FDC tablet orally once daily for 12 weeks in participants with genotype 2 (GT-2) HCV infection
- SOF/VEL (GT-3): SOF/VEL (400/100 mg) FDC tablet orally once daily for 12 weeks in participants with genotype 3 (GT-3) HCV infection
- SOF/VEL (GT-4): SOF/VEL (400/100 mg) FDC tablet orally once daily for 12 weeks in participants with genotype 4 (GT-4) HCV infection
- SOF/VEL (GT-6): SOF/VEL (400/100 mg) FDC tablet orally once daily for 12 weeks in participants with genotype 6 (GT-6) HCV infection
- SOF/VEL (Indeterminate): SOF/VEL (400/100 mg) FDC tablet orally once daily for 12 weeks in participants with indeterminate genotype HCV infection
- Total: Total of all reporting groups
Arm/Group | SOF/VEL (GT-1) | SOF/VEL (GT-2) | SOF/VEL (GT-3) | SOF/VEL (GT-4) | SOF/VEL (GT-6) | SOF/VEL (Indeterminate) | Total
Number analyzed (Participants) | 25 | 7 | 16 | 4 | 2 | 5 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (11.9) | 67 (13.5) | 55 (8.4) | 58 (15.5) | 69 (3.5) | 52 (13.0) | 60 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 4 | 5 | 1 | 1 | 3 | 24
  Male | 15 | 3 | 11 | 3 | 1 | 2 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 0 | 0 | 1 | 3
  Not Hispanic or Latino | 23 | 7 | 16 | 4 | 2 | 4 | 56
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Asian | 6 | 1 | 7 | 1 | 2 | 1 | 18
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Black or African American | 1 | 2 | 0 | 2 | 0 | 1 | 6
  White | 16 | 4 | 7 | 1 | 0 | 3 | 31
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
IL28b Status [Count of Participants; unit: Participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  Participants
    CC | 9 | 4 | 6 | 0 | 1 | 3 | 23
    CT | 14 | 1 | 8 | 4 | 1 | 2 | 30
    TT | 2 | 2 | 2 | 0 | 0 | 0 | 6
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.0 (0.70) | 5.2 (1.04) | 6.4 (0.55) | 5.6 (1.55) | 6.4 (0.27) | 4.4 (1.69) | 5.8 (1.02)
HCV RNA Category [Count of Participants; unit: Participants]
  < 800,000 IU/mL | 12 | 5 | 4 | 2 | 0 | 3 | 26
  ≥ 800,000 IU/mL | 13 | 2 | 12 | 2 | 2 | 2 | 33

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 15 IU/mL) 12 weeks after stopping the study treatment.
Time Frame: Posttreatment Week 12
Population: The Full Analysis Set included participants who are enrolled into the study and received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- SOF/VEL (Total): SOF/VEL (400/100 mg) FDC tablet orally once daily for 12 weeks
Arm/Group | SOF/VEL (Total) | SOF/VEL (GT-1) | SOF/VEL (GT-2) | SOF/VEL (GT-3) | SOF/VEL (GT-4) | SOF/VEL (GT-6) | SOF/VEL (Indeterminate)
Number analyzed (Participants) | 59 | 25 | 7 | 16 | 4 | 2 | 5
percentage of participants | 94.9 [85.9 to 98.9] | 92.0 [74.0 to 99.0] | 100.0 [59.0 to 100.0] | 93.8 [69.8 to 99.8] | 100.0 [39.8 to 100.0] | 100.0 [15.8 to 100.0] | 100.0 [47.8 to 100.0]

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued the Study Drug Due to an Adverse Event
Time Frame: First dose date up to Week 12
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- SOF/VEL: SOF/VEL (400/100 mg) FDC tablet orally once daily for 12 weeks
Arm/Group | SOF/VEL
Number analyzed (Participants) | 59
percentage of participants | 0

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 4 Weeks After Discontinuation of Therapy (SVR4)
Description: SVR4 was defined as HCV RNA < LLOQ 4 weeks after stopping study treatment.
Time Frame: Posttreatment Week 4
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL (Total) | SOF/VEL (GT-1) | SOF/VEL (GT-2) | SOF/VEL (GT-3) | SOF/VEL (GT-4) | SOF/VEL (GT-6) | SOF/VEL (Indeterminate)
Number analyzed (Participants) | 59 | 25 | 7 | 16 | 4 | 2 | 5
percentage of participants | 96.6 [88.3 to 99.6] | 96.0 [79.6 to 99.9] | 100.0 [59.0 to 100.0] | 93.8 [69.8 to 99.8] | 100.0 [39.8 to 100.0] | 100.0 [15.8 to 100.0] | 100.0 [47.8 to 100.0]

4. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 24 Weeks After Discontinuation of Therapy (SVR24)
Description: SVR24 was defined as HCV RNA < LLOQ 24 weeks after stopping study treatment.
Time Frame: Posttreatment Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL (Total) | SOF/VEL (GT-1) | SOF/VEL (GT-2) | SOF/VEL (GT-3) | SOF/VEL (GT-4) | SOF/VEL (GT-6) | SOF/VEL (Indeterminate)
Number analyzed (Participants) | 59 | 25 | 7 | 16 | 4 | 2 | 5
percentage of participants | 94.9 [85.9 to 98.9] | 92.0 [74.0 to 99.0] | 100.0 [59.0 to 100.0] | 93.8 [69.8 to 99.8] | 100.0 [39.8 to 100.0] | 100.0 [15.8 to 100.0] | 100.0 [47.8 to 100.0]

5. Secondary Outcome: Change From Baseline in HCV RNA
Time Frame: Baseline; Weeks 2, 4, 6, 8, and 12
Population: Participants in the Full Analysis Set with available date were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL (Total) | SOF/VEL (GT-1) | SOF/VEL (GT-2) | SOF/VEL (GT-3) | SOF/VEL (GT-4) | SOF/VEL (GT-6) | SOF/VEL (Indeterminate)
Number analyzed (Participants) | 59 | 25 | 7 | 16 | 4 | 2 | 5
log10 IU/mL
  Change at Week 2: number analyzed (Participants) | 55 | 25 | 6 | 13 | 4 | 2 | 5
  Change at Week 2 | -4.54 (1.017) | -4.69 (0.797) | -3.78 (0.840) | -5.07 (0.493) | -4.23 (1.333) | -5.29 (0.269) | -3.24 (1.668)
  Change at Week 4 | -4.69 (1.020) | -4.81 (0.704) | -4.05 (1.041) | -5.20 (0.551) | -4.48 (1.547) | -5.29 (0.269) | -3.26 (1.692)
  Change at Week 6 | -4.69 (1.020) | -4.81 (0.704) | -4.05 (1.041) | -5.20 (0.551) | -4.48 (1.547) | -5.29 (0.269) | -3.26 (1.692)
  Change at Week 8 | -4.69 (1.020) | -4.81 (0.704) | -4.05 (1.041) | -5.20 (0.551) | -4.48 (1.547) | -5.29 (0.269) | -3.26 (1.692)
  Change at Week 12 | -4.69 (1.020) | -4.81 (0.704) | -4.05 (1.041) | -5.20 (0.551) | -4.48 (1.547) | -5.29 (0.269) | -3.26 (1.692)

6. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ on Treatment
Time Frame: Weeks 2, 4, 6, 8, and 12
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL (Total) | SOF/VEL (GT-1) | SOF/VEL (GT-2) | SOF/VEL (GT-3) | SOF/VEL (GT-4) | SOF/VEL (GT-6) | SOF/VEL (Indeterminate)
Number analyzed (Participants) | 59 | 25 | 7 | 16 | 4 | 2 | 5
percentage of participants
  Week 2 | 67.8 [54.4 to 79.4] | 76.0 [54.9 to 90.6] | 85.7 [42.1 to 99.6] | 43.8 [19.8 to 70.1] | 50.0 [6.8 to 93.2] | 100.0 [15.8 to 100.0] | 80.0 [28.4 to 99.5]
  Week 4 | 100.0 [93.9 to 100.0] | 100.0 [86.3 to 100.0] | 100.0 [59.0 to 100.0] | 100.0 [79.4 to 100.0] | 100.0 [39.8 to 100.0] | 100.0 [15.8 to 100.0] | 100.0 [47.8 to 100.0]
  Week 6 | 100.0 [93.9 to 100.0] | 100.0 [86.3 to 100.0] | 100.0 [59.0 to 100.0] | 100.0 [79.4 to 100.0] | 100.0 [39.8 to 100.0] | 100.0 [15.8 to 100.0] | 100.0 [47.8 to 100.0]
  Week 8 | 100.0 [93.9 to 100.0] | 100.0 [86.3 to 100.0] | 100.0 [59.0 to 100.0] | 100.0 [79.4 to 100.0] | 100.0 [39.8 to 100.0] | 100.0 [15.8 to 100.0] | 100.0 [47.8 to 100.0]
  Week 12 | 100.0 [93.9 to 100.0] | 100.0 [86.3 to 100.0] | 100.0 [59.0 to 100.0] | 100.0 [79.4 to 100.0] | 100.0 [39.8 to 100.0] | 100.0 [15.8 to 100.0] | 100.0 [47.8 to 100.0]

7. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as:
  * On-treatment virologic failure:
    * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
    * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
    * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
  * Virologic relapse:
    * Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit
Time Frame: Baseline to Posttreatment Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL (Total) | SOF/VEL (GT-1) | SOF/VEL (GT-2) | SOF/VEL (GT-3) | SOF/VEL (GT-4) | SOF/VEL (GT-6) | SOF/VEL (Indeterminate)
Number analyzed (Participants) | 59 | 25 | 7 | 16 | 4 | 2 | 5
percentage of participants | 3.4 | 4.0 | 0 | 6.3 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants Who Develop Viral Resistance (as Assessed by Presence of HCV NS5A and NS5B Genes) to SOF and VEL During Treatment and After Discontinuation of Treatment
Description: Baseline deep sequencing of the HCV NS5A and NS5B genes was performed for all participants. For all participants with virologic failure, deep sequencing was performed at the first time point after virologic failure if the plasma or serum sample was available and HCV RNA was > 1000 IU/mL.
Time Frame: First dose date up to Posttreatment Week 24
Population: Participants in the Resistance Analysis Population Set included all participants in the Safety Analysis Set with a virologic outcome and at least 1 gene sequenced. All data are reported at a 15% assay cutoff.
Measure: Count of Participants; unit: Participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 58
Participants | 0

9. Secondary Outcome: Pharmacokinetic (PK) Parameter: AUCtau of SOF
Description: AUCtau is defined as the population PK derived area under the concentration versus time curve of the drug over the dosing interval.
Time Frame: Sparse PK samples at Weeks 6, 8, and 12 (all participants). Intensive PK samples at predose, 0.25, 0.5, 1, 2, 4, 6, 8, 10, and 12 hours postdose once at Week 6, 8, or 12 (participants who enrolled in the optional PK substudy (N=1))
Population: Participants in the PK Analysis Set (all participants who took at least 1 dose of study drug and had at least 1 nonmissing postdose concentration value for the corresponding analyte in plasma) with available data were analyzed. Population PK analyses of all sparse and intensive PK data were utilized to estimate steady-state AUCtau of SOF.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | SOF/VEL
Number analyzed (Participants) | 21
h*ng/mL | 2381.9 (567.63)

10. Secondary Outcome: PK Parameter: AUCtau of GS-331007 (Metabolite of SOF)
Description: as for outcome 9
Time Frame: as for outcome 9
Population: Participants in the PK analysis Set were analyzed. Population PK analyses of all sparse and intensive PK data were utilized to estimate steady-state AUCtau of GS-331007 .
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | SOF/VEL
Number analyzed (Participants) | 59
h*ng/mL | 230989.2 (81453.30)

11. Secondary Outcome: PK Parameter: AUCtau of VEL
Description: AUCtau is defined as the population PK derived area under the concentration verses time curve of the drug over the dosing interval.
Time Frame: as for outcome 9
Population: Participants in the PK Analysis Set were analyzed. Population PK analyses of all sparse and intensive PK data were utilized to estimate steady-state AUCtau of VEL.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | SOF/VEL
Number analyzed (Participants) | 59
h*ng/mL | 4279.4 (2198.77)

12. Secondary Outcome: PK Parameter: Cmax of SOF
Description: Cmax is defined as the population PK derived maximum concentration of the drug.
Time Frame: as for outcome 9
Population: Participants in the PK Analysis set with available data were analyzed. Population PK analyses of all sparse and intensive PK data were utilized to estimate steady-state Cmax of SOF.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SOF/VEL
Number analyzed (Participants) | 21
ng/mL | 1041.0 (176.96)

13. Secondary Outcome: PK Parameter: Cmax of GS-331007 (Metabolite of SOF)
Description: Cmax is defined as the population PK derived maximum concentration of the drug.
Time Frame: as for outcome 9
Population: Participants in the PK Analysis Set were analyzed. Population PK analyses of all sparse and intensive PK data were utilized to estimate steady-state Cmax of GS-331007.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SOF/VEL
Number analyzed (Participants) | 59
ng/mL | 9776.2 (3433.16)

14. Secondary Outcome: PK Parameter: Cmax of VEL
Description: Cmax is defined as the population PK derived maximum concentration of the drug.
Time Frame: as for outcome 9
Population: Participants in the PK Analysis Set were analyzed. Population PK analyses of all sparse and intensive PK data were utilized to estimate steady-state Cmax of VEL.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SOF/VEL
Number analyzed (Participants) | 59
ng/mL | 226.9 (92.80)

15. Secondary Outcome: PK Parameter: Ctau of VEL
Description: Ctau is defined as the population PK derived concentration of the drug at the end of a 24 hour dosing interval. The 24 hour Ctau is estimated based on the combination of sparse PK samples collected at random times across the dosing interval as well as intensive PK samples collected for up to 12 hours post-dose.
Time Frame: as for outcome 9
Population: Participants in the PK Analysis Set were analyzed. Population PK analyses of all sparse and intensive PK data were utilized to estimate steady-state Ctau of VEL.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SOF/VEL
Number analyzed (Participants) | 59
ng/mL | 137.2 (95.91)

ADVERSE EVENTS:
Time Frame: Adverse Events: First dose date up to Week 12 plus 30 days; All-Cause Mortality: First dose date up to Posttreatment Week 24
Description: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Arm/Group | SOF/VEL
All-Cause Mortality (participants affected / at risk) | 2/59
Serious Adverse Events (participants affected / at risk) | 11/59
Other Adverse Events (participants affected / at risk) | 33/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL (N=59)
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Cellulitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Lower respiratory tract infection viral (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Streptococcal bacteraemia (Infections and infestations) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Post procedural swelling (Injury, poisoning and procedural complications) | 1
Pubis fracture (Injury, poisoning and procedural complications) | 1
Neurilemmoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL (N=59)
Constipation (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 8
Fatigue (General disorders) | 8
Decreased appetite (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 5
Headache (Nervous system disorders) | 10
Insomnia (Psychiatric disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2017-03-02): https://cdn.clinicaltrials.gov/large-docs/52/NCT03036852/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-05): https://cdn.clinicaltrials.gov/large-docs/52/NCT03036852/SAP_001.pdf